CLINICAL TRIAL: NCT05579028
Title: Prospective Open-label Comparative in Two-group Investigator-initiated Low-interventional Study to Assess the Effect of Oral Nutritional Supplement (ONS) Nutridrink® 200 ml on the Ability of Patients With COVID-19 to Health Recovery
Brief Title: Study to Assess the Effect of ONS Nutridrink® 200 ml on the Recovery of Patients With COVID-19 and Respiratory Support
Status: Completed | Type: Observational
Sponsor: Enrollme.ru, LLC (Network)
Collaborators: Danone Nutricia (Industry)
Responsible Party: Sponsor
Other Study IDs: RECOVID
Record Dates: First submitted 2022-10-12; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
Keywords: covid-19; ICU; respiratory support; quality of life; physical recovery
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study: Patients of the group received supplemental nutritional support with Nutridrink ONS 200 ml, 2 bottles (400 ml) daily for 28 days from the date of inclusion. In a hospital setting, additional nutritional support will be added to the patient's standard hospital diet. After being discharged from the hospital, the patient will receive at his disposal the required amount of Nutridrink ONS 200 ml in amount of 400 ml per day and will take it in addition to his usual and habitual diet. The Nutridrink ONS 200 ml is recommended to be taken between main meals.
  Interventions: Dietary Supplement: Nutridrink ONS 200 ml
- Control: Patients of the group received a standard hospital diet, and upon discharge from the hospital - their usual habitual diet.

INTERVENTIONS:
Dietary Supplement: Nutridrink ONS 200 ml — Nutridrink is a high-protein, high-calorie formula for the specialized nutrition of patients with or at risk of malnutrition. The product can be used as an additional or sole source of nutrition
  Groups: Study

SUMMARY:
The goal of this low-interventional study was to learn about the effect a nutritional supplement in patients with COVID-19 and respiratory support. The main questions it aimed to answer were:

* if additional nutrition support has an effect on recovery of physical health in patients with COVID-19;
* to examine the effect of additional nutrition support on quality of life of patients with COVID-19;
* to examine the effect of the additional nutrition support on hospitalization period of patients with COVID-19.

Participants were split into two groups. One group had the common hospital diet, another group in addition to the common diet was given with NutriDrink® 200 ml X 2 daily. During the observation period participants were asked to measure hand strength measured by hand grip tester and fill out the quality of life standard questionnaire SF-36. In addition, several routine blood tests were performed.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed new coronavirus infection COVID-19 (based on laboratory and/or computer tomography data);
* Need in respiratory support (oxygen insufflation, non-invasive lung ventilation, artificial lung ventilation, as well in a prone position);
* Ability to take food spontaneously in the amount of 60% and more of energy and protein needs (possibility of spontaneous food intake will be determined with the three-swallow test; consumed food will be controlled with the "quarter of a plate" method);
* The informed consent is signed by a patient for the study enrollment and processing of personal data.

Exclusion Criteria:

* Diabetes mellitus;
* Renal failure;
* Hepatic failure;
* Systemic disease;
* Active cancer;
* Poor survival prognosis.
* Aggravation of a patient's condition requiring his transfer to enteral feeding and/or parenteral nutrition;
* Occurrence of complications requiring surgical interventions;
* Patient's transfer for treatment to another inpatient unit;
* Complications induced by the product for additional nutrition support (diarrhea, nausea, vomiting);
* Withdrawal of the informed consent for the study enrollment and processing of personal data.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 185 patients infected with a new coronavirus infection COVID-19 and getting respiratory support were enrolled to the study in accordance with the inclusion/exclusion criteria. Patients were randomly devided into two groups.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Quality of life score, part "Physical Health component" according to the SF-36 questionnaire | up to 4 weeks
  SF-36 questionnaire
Quality of life score, part "Mental Health component" according to the SF-36 questionnaire | up to 4 weeks
  SF-36 questionnaire
Quality of life score "Total Quality of Life" according to the SF-36 questionnaire | up to 4 weeks
  SF-36 questionnaire
Change in handgrip (decanewton) strength between visits 3 and 1 | between inclusion and discharge from hospital (about 2-3 weeks)
  Hand grip measured with hand dynamometer

SECONDARY OUTCOMES:
Duration (days) of the patient stay under respiratory support or in the intensive care unit | during observation
  Medical record
Total stay in the hospital (days) | during observation
  Medical record
Severity of the current status according to the Post-COVID19 Functional Status (PCFS) Scale | during observation
  PCFS is not validated but usefull tool to measure patients' functional status https://erj.ersjournals.com/content/56/1/2001494
Nutritional Impact Symptom (NIS) Check-list score | during observation
  check-list and scale developed for cachexia patients and published in https://link.springer.com/article/10.1007/s13539-012-0099-x

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail A Getman, Dr, Study Director — Enrollme.ru
Locations (6):
- Russia (6):
  - City clinical hospital # 4, Moscow
  - Pirogov Medical university, Moscow
  - City clinical hospital # 11, Omsk
  - City clinical hospital by Saint George the Great Martyr, Saint Petersburg
  - Pokrovskaya hospital, Saint Petersburg
  - Central city clinical hospital # 24, Yekaterinburg